CLINICAL TRIAL: NCT00632606
Title: Magnesium Sulfate vs Metoclopramide for Headache in Pregnant Women
Brief Title: MgSO4 vs Metoclopramide for Headache in Pregnant Women
Acronym: MagHead
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Ghada Bourjeily, Dr. Ghada Bourheily, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB#08-0006
Record Dates: First submitted 2008-02-29; First posted 2008-03-11 (Estimated); Last update posted 2012-12-25 (Estimated); Status verified 2012-12

CONDITIONS: Headache
Keywords: pregnant women
MeSH Terms: conditions — Headache | interventions — Magnesium Sulfate; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): magnesium sulfate 2 grams intravenously w/ acetaminophen 1 gram orally
  Interventions: Drug: magnesium sulfate
- Arm 2 (Active Comparator): metoclopramide 10 mg intravenously w/ 1 gram acetominophen orally
  Interventions: Drug: metoclopramide

INTERVENTIONS:
Drug: magnesium sulfate — magnesium sulfate 2 grams intravenously; both groups will receive acetaminophen (Tylenol®) 1 gram orally
  Arms: Arm 1
Drug: metoclopramide — metoclopramide 10 mg intravenously; both groups will receive acetaminophen (Tylenol®) 1 gram orally
  Other Names: Reglan
  Arms: Arm 2

SUMMARY:
The study will compare effectiveness of intravenous magnesium sulfate to that of intravenous metoclopramide (Reglan®) for acute headache in pregnant women. We will randomize pregnant women who present to our emergency department with chief complaint of headache to magnesium sulfate 2 grams intravenously or metoclopramide 10 mg intravenously; both groups will receive acetaminophen (Tylenol®) 1 gram orally and normal saline 1 liter intravenously. Headaches are common during pregnancy, related to hormonal changes, altered sleep patterns and psychosocial stressors. Common medications for headache such as non-steroidal antiinflammatories or triptans are typically avoided during pregnancy due to concern for fetal effects. Women, and their physicians, are often uncertain regarding available medication options with justifiable safety profiles during pregnancy.

DETAILED DESCRIPTION:
Metoclopramide and prochlorperazine (Compazine®), antiemetic dopamine receptor antagonists, are widely used for headache treatment in North American emergency departments. Metoclopramide, FDA pregnancy category B, is used in clinical practice for acute headache in pregnant women. Small studies have found magnesium sulfate to be effective in migraine, tension and cluster headaches, although there is no data regarding efficacy or tolerability in pregnant women.

Our study would be similar to a Turkish study published in 2004 which compared magnesium sulfate to metoclopramide for acute headache treatment in nonpregnant individuals; they found the drugs equally effective 30 minutes after administration. Serum magnesium levels in pregnant women are often lower than in nonpregnant women; magnesium deficiency has been explored as contributing to headache frequency and severity. Magnesium sulfate use has been well established during pregnancy for decades, administered intravenously to delay labor or to women with preeclampsia for 24 to 48 hours, initially with 4 to 6 gram bolus then 2 grams per hour. For headache treatment, magnesium sulfate dose would be far lower, 2 grams. We would like to determine the efficacy and tolerability of magnesium sulfate for headache relief in pregnant women, as well as evaluate efficacy of metoclopramide in pregnant women. We do not find published randomized trials evaluating headache treatment in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant, 18-75
* Headache rated 4 or greater on a 0-10 pain scale

Exclusion Criteria:

* New objective neurologic abnormality at the time of exam
* Temperature >100.4
* Allergy or intolerance to study medications
* Suspected of confirmed preeclampsia/eclampsia
* Complete heart block
* Hypotension, SBP<85
* Myasthenia gravis
* End stage renal failure

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The study will compare effectiveness of intravenous magnesium sulfate to that of intravenous metoclopramide (Reglan®) for acute headache in pregnant women. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Hayes, MD, Principal Investigator — Women and Infants Hospital of Rhode Island
Locations (1):
- Women and Infants Hospital of Rhode Island, Providence, Rhode Island, United States